CLINICAL TRIAL: NCT06943807
Title: Research on the Application of Fecal DNA Methylation Detection in the Early Diagnosis and Screening of Gastric Cancer
Brief Title: Fecal DNA Methylation Detection for Gastric Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Director, Fudan University
Other Study IDs: 2014-Exp079
Record Dates: First submitted 2025-03-17; First posted 2025-04-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Fecal sample methylation detection for gastric cancer — Detection of gastric cancer-associated methylation sites in fecal samples

SUMMARY:
The study is a prospective, multicentre, cross-sectional study to evaluate the efficacy of fecal methylation-based testing in comparison with the 'gold standard' imaging tests, such as CT, gastroscopy and/or pathology, for the prediction of gastric cancer in an enrolled population.

DETAILED DESCRIPTION:
Aims of the study Primary study aim: To assess the sensitivity and specificity of fecal methylation site-based tests for the prediction of gastric cancer.

Secondary research objectives: 1. the accuracy, kappa value, area under the ROC curve, positive likelihood ratio, negative likelihood ratio, positive predictive value, negative predictive value of fecal methylation locus test for the prediction of gastric cancer; 2. whether the predictive ability is significantly higher than that of conventional tumour markers, such as CA19-9, CEA, and CA72-4, etc.; 3. The predictive ability of the combined fecal H. pylori gastric cancer susceptibility test was assessed.

Study design Prospective, multicentre, cross-sectional study. Study period 2 years from the start of the project as approved by the Institutional Ethics Committee.

Target population The target population is over 40 years old in areas with a high incidence of gastric cancer.

Sample size The sample size of this study should not be less than 10,800 cases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years, male or female.
* Have or will have gastroscopy and/or pathology results.
* No contraindications to endoscopy and able to cooperate with endoscopy.
* Patients must be able to fully understand the informed consent form and be able to sign the informed consent form in person.

Exclusion Criteria:

* Have severe cardiac, hepatic, or renal insufficiency, or mental disorders.
* Previous history of upper gastrointestinal malignancy.
* Women during pregnancy.
* Those with unspecified pathology.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this clinical study were obtained from inpatients and outpatient follow-up patients attending the two sub-centers. Subjects were identified by the investigator based on subject enrollment criteria and informed of the contents of the informed consent form.
Sampling Method: Probability Sample
Enrollment: 10800 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of fecal DNA methylation testing based on its application for early diagnosis and screening of gastric cancer. | Baseline

IPD SHARING:
Plan to Share IPD: Undecided